CLINICAL TRIAL: NCT03165227
Title: Randomised, Double-blind, Placebo-controlled Trial to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of 3 Multiple Rising Oral Doses of BI 685509 Over 28 Days in Male and Female Patients With Diabetic Nephropathy
Brief Title: This Study Tests a New Medicine Called BI 685509 in Patients That Have Kidney Problems Because of Diabetes. The Study Tests How BI 685509 is Taken up in the Body and How Well it is Tolerated (Multiple Rising Doses)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 1366-0004; 2014-004541-27 (EudraCT Number)
Record Dates: First submitted 2017-05-23; First posted 2017-05-24 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Diabetic Nephropathies
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BI 685509 Dose 1 (Experimental)
  Interventions: Drug: BI 685509
- BI 685509 Dose 2 (Experimental)
  Interventions: Drug: BI 685509
- BI 685509 Dose 3 (Experimental)
  Interventions: Drug: BI 685509
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 685509 — Taken orally
  Arms: BI 685509 Dose 1; BI 685509 Dose 2; BI 685509 Dose 3
Drug: Placebo — Taken orally
  Arms: Placebo

SUMMARY:
The main objective of this trial is the safety and tolerability of 3 multiple rising oral doses of BI 685509 over 28 days in male and female patients with Diabetic Nephropathy (DN) as adjunctive to Angiotensin Converting Enzyme inhibitor (ACEi) or Angiotensin Receptor Blocker (ARB). Another objective is the change in Urine Albumin Creatinine Ratio (UACR), an important diagnostic marker of nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial
* Male or postmenopausal (last menstruation ≥ 2 years ago) patients, or female patients who are sterilized by either hysterectomy, bilateral salpingectomy and/or bilateral oophorectomy. Male patients with partners of child-bearing potential must be willing to use condoms from the time of the first intake of study drug until follow-up.
* eGFR (Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula) ≥ 20 and < 75 ml/min/1.73 m2 at Visit 1 measured by the central laboratory and no planned start of renal replacement therapy during the trial
* UACR ≥ 200 and <3500 mg/g in spot urine (midstream urine sample) at Visit 1 measured by the central laboratory
* Treatment with either ACEi or ARB, stable dose since ≥ 4 weeks before Visit 1 with no planned change of the therapy
* Patients with type 1 or type 2 diabetes mellitus, diagnosed before informed consent and treated with insulin, glucagon-like peptide (GLP) 1 agonists and/or oral antidiabetic medication. Treatment should have been unchanged (investigator's judgment) within 4 weeks before Visit 1 and until randomisation
* Glycated Haemoglobin (HbA1c) < 10.0% at Visit 1 measured by the central laboratory
* Seated Systolic Blood Pressure (SBP) ≥ 110 and ≤ 180 mmHg and Diastolic Blood Pressure (DBP) ≥ 70 and ≤ 110 mmHg at Visit 1
* Age at screening ≥ 18 years for male and permanently sterilized female patients and ≥ 45 years for postmenopausal female patients
* Body Mass Index (BMI) ≥ 18.5 and < 45 kg/m2
* Successful ABPM reading before randomisation, upper arm circumference within the circumference level of the cuff size of either ABPM and/or BP measurement device used in the study

Exclusion Criteria:

* Treatment with SGLT2 inhibitors and/or phosphodiesterase inhibitors, nitrates or riociguat, from screening (Visit 1) or within 5 half-lives before randomisation whatever is earlier.
* Any laboratory value more than 3 times above upper limit of normal (ULN) at screening (Visit 1) or any other laboratory value outside the reference range and clinically relevant (for safe participation) in the investigator judgment
* Confirmed non-diabetic renal disease in the opinion of investigator
* Any other medical condition that in the investigator's opinion poses a safety risk for the patient or may interfere with the study objectives including

  * symptomatic heart failure (NYHA III/IV),
  * known history of tachycardia and/or atrial fibrillation
  * clinically relevant arrhythmias
  * coronary heart disease not compensated by medical treatment (supine pulse rate >70 beats per minute, existing angina pectoris)
  * <6 months after myocardial infarction.
* Medical history of cancer or treatment for cancer in the last two years prior to Visit 1 (except appropriately treated basal cell carcinoma of the skin, in situ carcinoma of uterine cervix, and prostatic cancer of low grade [T1 or T2] is exempted)
* Surgery or trauma with significant blood loss (investigator's judgement) within the last 3 months prior to informed consent or significant blood donation (investigator's judgement) within four weeks prior to first administration of study medication or planned during the trial
* Previous randomization in this trial
* Currently enrolled in another investigational device or drug study, i.e., less than 30 days since ending another investigational device or drug study(s), or receiving other investigational treatment(s)
* Chronic alcohol or drug abuse or any condition that, in the investigator's opinion, makes them an unreliable study subject or unlikely to complete the trial
* Women of childbearing potential
* Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with drug related Adverse Events (AEs) | Up to 35 days

SECONDARY OUTCOMES:
Change from baseline in log transformed Urine albumin creatinine ratio (UACR) measured in morning void urine | Up to 28 days
Change from baseline in log transformed Urine albumin creatinine ratio (UACR) measured in 10-hour urine | Up to 28 days

CONTACTS AND LOCATIONS:
Locations (35):
- United States (22):
  - Nephrology Consultants, LLC, Huntsville, Alabama
  - California Institute of Renal Research, La Mesa, California
  - Office of Dr. Richard S. Cherlin, Los Gatos, California
  - Creekside Endocrine Associates, PC, Denver, Colorado
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - The Center for Diabetes and Endocrine Care, Fort Lauderdale, Florida
  - Indago Research and Health Center, Hialeah, Florida
  - South Florida Research Institute, Lauderdale Lakes, Florida
  - San Marcus Research Clinic, Inc., Miami, Florida
  - Ocean Blue Medical Research Center, Inc., Miami Springs, Florida
  - Genesis Clinical Research, Tampa, Florida
  - Boise Kidney and Hypertension Institute, Meridian, Idaho
  - Research by Design, LLC, Chicago, Illinois
  - Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Northwest Louisiana Nephrology L.L.C., Shreveport, Louisiana
  - Scott Research, Inc., Laurelton, New York
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Knoxville Kidney Center PLLC, Knoxville, Tennessee
  - Research Institute of Dallas, Dallas, Texas
  - Houston Clinical Research Associates, Houston, Texas
  - Science Advancing Medicine Clinical Research Center, San Antonio, Texas
  - York Clinical Research, LLC, Norfolk, Virginia
- Belgium (5):
  - Bonheiden - HOSP Imelda, Bonheiden
  - Brussels - UNIV UZ Brussel, Brussels
  - Edegem - UNIV UZ Antwerpen, Edegem
  - UNIV UZ Gent, Ghent
  - Centre Hospitalier Universitaire de Liège, Liège
- Toronto General Hospital, Toronto, Ontario, Canada
- Czechia (5):
  - University Hospital Brno, Brno
  - St. Anna Hospital, 2nd Internal Department, Brno
  - Quinta Analytica, Prague
  - Institute for Clinical and Experimental Medicine, Prague
  - General University Hospital in Prague, Prague
- Germany (2):
  - SocraTec R&D GmbH, Erfurt
  - CTC North GmbH & Co. KG, Hamburg, Hamburg